CLINICAL TRIAL: NCT04731636
Title: Guo's Visceral Arteries Reconstruction :The First in Man Study of G-Branch Multiple Branch Stent Graft System.
Brief Title: Guo's Visceral Arteries Reconstruction: First in Man Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, XuWei, Project manager, Lifetech Scientific (Shenzhen) Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAAA-FIM-001
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Pararenal Aortic Aneurysm
Keywords: Guo's Visceral Arteries Reconstruction; Thoracoabdominal aortic stent system; Thoracoabdominal Aortic Aneurysms; G-Branch; Pararenal abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- G-Branch Thoracoabdominal Aortic Stent System (Experimental): Patients with Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm, and passed the screening and signed the Informed Consent Form
  Interventions: Device: Thoracoabdominal aortic stent system

INTERVENTIONS:
Device: Thoracoabdominal aortic stent system — Patients who meet all inclusion criteria and don't meet any exclusion criteria were implanted with thoracoabdominal aortic stent system.

SUMMARY:
A First in man study to evaluate the safety and efficacy of thoracoabdominal aortic stent system for thoracoabdominal aortic aneurysms and pararenal abdominal aortic aneurysm.

DETAILED DESCRIPTION:
The study is mainly for patients with Crawford type I-V thoracoabdominal aortic aneurysms and pararenal abdominal aortic aneurysm, and all subjects who passed the screening and signed the informed consent will be enrolled. Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with thoracoabdominal aortic stent system.

Patients will be followed up at discharge, 1 month, 6 months, 12 months after the implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years;
2. Patients diagnosed with type Crawford I-V thoracoabdominal aortic aneurysmsa and pararenal abdominal aortic aneurysm, and should meet at least one of the following conditions:

   1. The maximum diameter of thoracoabdominal aortic aneurysms and pararenal abdorminal aortic aneurysm > 50 mm;
   2. Rapid growth of sac >5 mm in diameter in the most recent 6 months;
   3. Definite symptoms of abdominal pain and low back pain associated with thoracicabdominal aortic aneurysms.
3. Patients with four indispensable reno-visceral arteries including superior mesenteric artery, celiac trunk and bilaterial renal arteries.
4. Proximal landing zone 20-36 mm in diameter;
5. Proximal landing zone ≥25 mm in length;
6. If distal landing zone in abdominal aorta, distal landing zone should be 12-36mm in diameter and ≥15 mm in length.
7. The visceral vascular branches landing zone 6~13 mm in diameter and ≥15 mm in length;
8. The renal artery landing zone 4.5~9 mm in diameter and ≥15 mm in length;
9. Patients who using the abdominal aortic bifurcation stent graft system should also meet the following criteria:

   1. The ilac artery landing zone 7 ~25 mm in diameter;
   2. The ilac artery landing zone ≥15 mm in length;
10. Patients with appropriate iliacofemoral access and at least one patent upper extremity access;
11. Patients who can understand the purpose of the trial, volunntarily participate and sign the informed consent form, and are willing to complete the follow-up according to the requirements of the protocol;

Exclusion Criteria:

1. Ruptured aortic aneurysm in unstable haemodynamic condition;
2. Aneurysmal aortic dissection;
3. Infected or mycotic aortic aneurysm;
4. Requiring simultaneous coverage or embolisation for bilateral internal iliac arteries;
5. Severe stenosis, calcification, or mural thrombus at stent-graft landing zone;
6. Diagnosis of acute coronary syndrome within 6 months;
7. Patients with any transient ischemic attack (TIA) or ischemic stroke within 3 months;
8. An allergic history for contrast agents, anticoagulants, antiplatelet drugs, stent graft or materials of delivery system；
9. Patients with connective tissue diseases;
10. Patients with takayasu arteritis;
11. Patients with serious vital organ dysfunction or other serious disease;
12. Preoperative liver renal function abnormalities (ALT or AST ≥ 5 times the upper limit of normal value), or serum creatinine ≥ 150 μmol/L;
13. Severe pulmonary insufficiency who cannot tolerate general anaesthesia;
14. Severe coagulation dysfunction;
15. Undergone major surgical or interventionic surgery within 30 days before surgery;
16. Patients whose systemic or local infection may increase the risk of intravascular graft infection;
17. Planning pregnancy, pregnancy, or breastfeeding;
18. The patient participated in other clinical trials or not completed or withdrawn from other clinical trials within the last 3 months at the time of screening period ;
19. Life expectancy less than 1 year;
20. Patients not appropriate for endovascular repair based on the investigators' clinical judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Professor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- G-Branch Thoracoabdominal Aortic Stent System: Patients with Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm, and passed the screening and signed the informed consent form.
  G-Branch thoracoabdominal aortic stent system: Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with thoracoabdominal aortic stent system.
Period: Overall Study
Arm/Group | G-Branch Thoracoabdominal Aortic Stent System
Started | 15 (Number of patients who treated for Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm with thoracoabdominal aortic stent system，meet all inclusion criteria and not meet any exclusion criteria and signed the Informed Consent Form)
Completed | 15 (Number of patients who had undergone repair of Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm using thoracoabdominal aortic stent system)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of patients who treated for Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm with thoracoabdominal aortic stent system，meet all inclusion criteria and not meet any exclusion criteria and signed the Informed Consent Form
Groups:
- G-Branch Thoracoabdominal Aortic Stent System: Patients with Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm, and passed the screening and signed the Informed Consent Form.
  G-Branch thoracoabdominal aortic stent system: Patients who meet all inclusion criteria and don't meet any exclusion criteria were implanted with thoracoabdominal aortic stent system.
Arm/Group | G-Branch Thoracoabdominal Aortic Stent System
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — presenting the age of the 15 enrolled patients as mean ± standard deviation (SD) with thoraco-abdominal or pararenal abdominal aortic aneurysm.
  years | 63.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex distribution of the enrolled 15 patients with thoraco-abdominal or pararenal abdominal aortic aneurysm
  Participants
    Female | 2
    Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of the 15 enrolled patients with thoraco-abdominal or pararenal abdominal aortic aneurysm (exclusively Chinese).
  Participants
    American Indian or Alaska Native | 0
    Asian | 15
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Region of the 15 enrolled patients with thoraco-abdominal or pararenal abdominal aortic aneurysm (exclusively from China).
  Participants
    China | 15
Society for Vascular Surgery(SVS) score [Median (Full Range); unit: units on a scale] — The SVS score ranges from 0 to 24 and comprises eight factors: Diabetes, Tobacco Use, Hypertension, Hyperlipemia, Cardiac Status, Carotid Disease, Renal Status, and Pulmonary Status. Each factor is scored individually, and the total score reflects the severity of the patient's condition, with higher values indicating a worse outcome.
  units on a scale | 6 [2 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE) Within 30 Days Postoperative
Description: Major Adverse events (MAE) are defined as all-cause death, liver failure, intestinal necrosis, splenic infarction, renal infarction, renal failure, cerebral infarction, paraplegia, myocardial infarction, and respiratory failure.
Time Frame: within 30-days postoperative
Population: Total number of cases available for evaluation of adverse events.
Measure: Number; unit: participants
Groups:
- G-Branch Thoracoabdominal Aortic Stent System: Patients with Crawford type I-V thoracoabdominal aortic aneurysms and Pararenal abdominal aortic aneurysm, and passed the screening and signed theInformed Consent Form.
  G-Branch thoracoabdominal aortic stent system: Patients who meet all the inclusion criteria and don't meet any exclusion criteria were planteded with thoracoabdominal aortic stent system.
Arm/Group | G-Branch Thoracoabdominal Aortic Stent System
Number analyzed (Participants) | 15
participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | G-Branch Thoracoabdominal Aortic Stent System
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Branch Thoracoabdominal Aortic Stent System (N=15)
Died of acute cerebral infarction (Vascular disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Branch Thoracoabdominal Aortic Stent System (N=15)
Minor type II endoleak (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT04731636/Prot_SAP_000.pdf